CLINICAL TRIAL: NCT03727282
Title: Use of Transtoracic Ecocargiogram With Calculation of Left Ventricular Volume Index in the Initial Adjustment of Initial Dose of Dobutamine in Patients With Heart Failure and Cardiogenic Shock
Brief Title: Left Ventricular Volume Index in the Adjustment of Initial Dose of Dobutamine in Heart Failure and Cardiogenic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-TAPSE
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Cardiogenic Shock; Heart Failure
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal strategy (Other): Initiate dobutamine at 5 mcg/kg/min and adjust dobutamine according to the attending physician
  Interventions: Procedure: adjust dobutamine according to the attending physician
- ejection volume index (Experimental): Initiate dobutamine at 5 mcg/kg/min and adjust dobutamine according to the ejection volume index
  Interventions: Procedure: adjust dobutamine according to the ejection volume index

INTERVENTIONS:
Procedure: adjust dobutamine according to the ejection volume index — adjust dobutamine dose
  Arms: ejection volume index
Procedure: adjust dobutamine according to the attending physician — adjust dobutamine dose
  Arms: Liberal strategy

SUMMARY:
Recent studies have suggested that the use of left ventricular ejection volume index calculation may aid in the hemodynamic management of critically ill patients. However, a prospective and randomized comparison in patients with heart failure for inotropic dose adjustment has not been described. The objective of this study was to evaluate the efficacy and safety of ejection volume index versus liberal strategy in adjusting dobutamine dose in patients with heart failure and low cardiac output. Methodology: A unicentric, randomized and prospective study will be performed in a comparative manner. Hospital data (test results, medical outcomes, dobutamine dose, complications) of patients will be analyzed for safety and effectiveness. Expected results: The use of ejection volume index is not inferior to the liberal strategy in the initial adjustment of the dose of dobutamine in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤ 40% documented on echocardiography
* BNP> 500 pg / mL
* Need for initiation of dobutamine and signs or symptoms of low cardiac output at admission defined by the presence of 2 or more of the following:

  * SBP ≤ 95 mmHg
  * FC> 100 bpm
  * Peripheral vasoconstriction,
  * Cold extremities,
  * Reference of decrease of urine output,
  * Nausea, vomiting and food intolerance,
  * Presence of organic dysfunction

Exclusion Criteria:

* Pregnancy.
* COPD
* Hepatical cirrhosis
* Atrioventricular block of 2nd or 3rd degree. and. SBP <80 mmHg or need for vasopressor.
* Use of definitive pacemaker.
* Body mass index greater than 40 kg / m2.
* Use of oral anticoagulant.
* Acute coronary syndrome.
* Indication of use of another inotropic other than dobutamine.
* Orotracheal intubation.
* Presence of significant pericardial effusion.
* Obstruction of left ventricular outflow tract.
* Serum creatinine> 5.0 mg / dL or hemodialysis.
* Presence of 2 or more clinical / laboratory / radiological criteria of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2020-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
base excess levels | 24 hours
  serum analysis
bicarbonate levels | 24 hours
  serum analysis
systolic and diastolic blood pressure | 24 hours
  physical evaluation
cardiac output | 24 hours
  echocardiography echocardiography
systolic volume | 24 hours
  echocardiography
urinary output | 24 hours
  urine analysis
arterial lactate levels | 24 hours
  serum analysis
central venous oxygen saturation levels | 24 hours
  serum analysis
BNP levels | 24 hours
  plasma analysis
troponin levels | 24 hours
  serum analysis
heart rate | 24 hours
  physical evaluation
creatinine levels | 24 hours
  serum analysis
urea levels | 24 hours
  serum analysis

SECONDARY OUTCOMES:
occurrence of sustained ventricular arrhythmia | 24 hours
  electrocardiography
need for orotracheal intubation | 24 hours
need for vasopressor or other inotropic association | 24 hours
  hipotension
need for mechanical circulatory assistance | 24 hours
lowering of consciousness level | 24 hours
  glasgow < 14
cardiorespiratory arrest | 24 hours
worsening of renal function | 24 hours
  increase 0.5 mg / dl in relation to admission creatinine
death | 24 hours
failure of dobutamine weaning up | 7 days
hospitalization time | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, MD, Principal Investigator — Unidade Clínica de Emergência